CLINICAL TRIAL: NCT00313092
Title: Does Plasma Matrix-metalloproteinase Activity Predict Glaucomas in Patients With OSAS (Obstructive Sleep Apnea Syndrome) and Does the Level of Plasma Matrix-metalloproteinase Activity Decrease After One Month of nCPAP-treatment
Brief Title: Obstructive Sleep Apnea Syndrome in Glaucoma
Status: Terminated | Type: Observational
Why Stopped: recruiting problems
Sponsor: Selim Orguel (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Selim Orguel, Prof. Dr., University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 045-LEJ-2004-002
Record Dates: First submitted 2006-04-10; First posted 2006-04-11 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Obstructive Sleep Apnea Syndrome; Glaucoma
Keywords: OSAS; glaucoma; MMP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: nCPAP treatment — treatment with positive air pressure during night

SUMMARY:
The aim of the study is to determine if plasma matrix-metalloproteinase activity can predict glaucoma in patients with OSAS and if the level of plasma matrix-metalloproteinase activity will decrease after one month of nCPAP-treatment.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of blindness world-wide. Chronic primary open-angle glaucoma is the most common form among Caucasian patients. The key feature of glaucoma is damage to the optic nerve head, which is not necessarily related to an increased intraocular pressure. The prevalence of glaucoma among the patients with sleep apnoea was 7,2%: normal-tension glaucoma 2,9%, primary open-angle glaucoma 4,3%. The prevalence of obstructive sleep apnoea syndrome (OSAS) is around 4-10% for men and 2-4% for women. Matrix metalloproteinases (MMPs) substrates include essentially all extracellular matrix components as well as a wide array of molecules involved in intracellular adhesion, cell-matrix interaction, and cell signalling. However, MMPs effects are not restricted to extracellular matrix degradation. The prevalence of increased MMP in patients with OSAS and its predicting value for an additional glaucoma are not known. Further, we do not know if treatment of OSAS with nasal continuous positive air pressure(nCPAP) can decrease the MMP activity. With this study, we want to determine the prevalence of MMP activity and the prevalence of glaucoma in patients with OSAS. Further, we want to investigate if a nCPAP treatment period of four weeks decreases the MMP activity.

ELIGIBILITY:
Inclusion Criteria:

* OSAS planned begin of a nCPAP treatment

Exclusion Criteria:

* Current malignancy
* Oral steroids

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sleep apnoe syndrom
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Eye Clinic Basel
Locations (1):
- University Hospital Basel, Eye Clinic, Basel, Canton of Basel-City, Switzerland